CLINICAL TRIAL: NCT01922245
Title: tDCS and Aphasia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Elizabeth Galletta, PhD, Assistant Professor, Hunter College of City University of New York
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 062951
Record Dates: First submitted 2013-08-02; First posted 2013-08-14 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Aphasia
Keywords: aphasia; therapy; stroke; language; naming; quality of life; tDCS; treatment
MeSH Terms: conditions — Aphasia; Stroke; Language

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anodal tDCS (Experimental): Soterix 1x1 device: anodal tDCS administered to the left hemisphere
  Interventions: Device: Soterix 1x1 tDCS

INTERVENTIONS:
Device: Soterix 1x1 tDCS — Anodal and sham tDCS will be administered. All of the participants will also receive behavioral speech-language therapy.

SUMMARY:
This project will investigate the use of noninvasive brain stimulation in the form of tDCS (transcranial direct current stimulation) in conjunction with speech-language therapy, for the improvement of language production in stroke survivors with aphasia. The hypothesis is that anodal tDCS and speech-language therapy will facilitate improved outcomes compared to speech therapy alone.

DETAILED DESCRIPTION:
Aphasia, commonly defined as impairment or loss of language functions, is a frequent and often chronic consequence of stroke, with detrimental effects on patient autonomy and health-related quality of life (HRQOL). Although beneficial in some cases, the effectiveness of behavioral therapy is often limited, and therefore new complementary treatments must be developed in order to improve rehabilitation of post-stroke aphasia.

In most individuals, language areas in the brain are localized in the left hemisphere. After stroke, there is evidence that the brain reorganizes such that either areas close to damaged language areas in the Left Hemisphere, or anatomically similar areas in the Right Hemisphere, are recruited to perform language tasks.

Recently, studies have begun to examine the effects of non-invasive brain stimulation on aphasia rehabilitation. One such technique is transcranial direct current stimulation (tDCS), which involves administering weak electrical currents through surface electrodes on the scalp. The effects can either stimulate an area, or inhibit an area of the brain. The main hypothesis is that stimulating language areas in the Left Hemisphere in conjunction with speech language therapy will facilitate reorganization of language-relevant areas of the brain, and improve expression.

The proposed study will compare the effects of transcranial direct current stimulation (tDCS) activating language centers in the Left Hemisphere and sham tDCS, in right-handed individuals with chronic post-stroke aphasia. This study will provide information on the effects of tDCS, in conjunction with speech-language therapy, on aphasia rehabilitation.

ELIGIBILITY:
Inclusion Criteria: single left hemisphere stroke, more than three months post stroke, right handed, no other medical problems, ages 18-100 -

Exclusion Criteria: more than one stroke, less than three months post stroke, other medical problems, pacemaker or other electronic implant (e.g. hip replacement), pregnancy

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change in naming performance in singles words and sentence context | change from baseline naming performance at two weeks and four weeks post treatment
  Naming will be tested using standardized tests such at the Boston Naming Test and or the Philadelphia Naming Test. In addition, sentence probes have been created that will assess naming in the sentence context throughout the study.

SECONDARY OUTCOMES:
change in sentence production | change from baseline performance at two weeks and four weeks post treatment
  Sentence production will be classified.
change in health related quality of life | change from baseline performance at two weeks and four weeks post treatment
  Scales of health related quality of life will be implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Galletta, PhD, Principal Investigator — Hunter College/City University of NY
Locations (1):
- Hunter College Brookdale Campus, New York, New York, United States

REFERENCES:
- [Background] Baker JM, Rorden C, Fridriksson J. Using transcranial direct-current stimulation to treat stroke patients with aphasia. Stroke. 2010 Jun;41(6):1229-36. doi: 10.1161/STROKEAHA.109.576785. Epub 2010 Apr 15. PMID 20395612
- [Background] Fiori V, Cipollari S, Di Paola M, Razzano C, Caltagirone C, Marangolo P. tDCS stimulation segregates words in the brain: evidence from aphasia. Front Hum Neurosci. 2013 Jun 14;7:269. doi: 10.3389/fnhum.2013.00269. eCollection 2013. PMID 23785323
- [Result] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving aphasia in patients after stroke. Cochrane Database Syst Rev. 2013 Jun 25;(6):CD009760. doi: 10.1002/14651858.CD009760.pub2. PMID 23799617